CLINICAL TRIAL: NCT04366947
Title: Comparison of Intraosseous Versus Intravenous Access in Suspected/Confirmed COVID-19 Patient in Prehospital Setting
Brief Title: Intravascular Access in Suspected/Confirmed COVID-19 Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lazarski University (Other)
Collaborators: Poznan University of Medical Sciences (Other); Medical University of Bialystok (Other); Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Assoc Prof PhD, Lazarski University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IO_PPE_1
Record Dates: First submitted 2020-04-23; First posted 2020-04-29 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Emergency Medicine; Cardiopulmonary Arrest; Shock
Keywords: intravascular access; intraosseous access; personal protective equipment; cardiopulmonary resuscitation; shock
MeSH Terms: conditions — Heart Arrest; Shock

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Intravenous Cannula) (Experimental): obtaining intravascular access using a ready standard intravenous cannula
  Interventions: Device: Standard of Care (Intravenous access)
- Experimental: IO access using NIO® set (Experimental): receive an IO line in the proximal tibia localization. IO lines are placed using an FDA-approved device called an NIO®.
  Interventions: Device: NIO® (Intraosseous access)

INTERVENTIONS:
Device: NIO® (Intraosseous access) — obtaining intravascular access using a ready intravenous NIO needle set
  Other Names: IO
  Arms: Experimental: IO access using NIO® set
Device: Standard of Care (Intravenous access) — obtaining intravascular access using a standard intravenous cannula
  Other Names: IV
  Arms: Standard of Care (Intravenous Cannula)

SUMMARY:
The current COVID-19 pandemic, this is especially since the transmission of SARS-CoV-2 is thought to occur mainly through respiratory droplets generated by coughing and sneezing, by direct contact with contaminated surfaces and because in a large number of patients COVID-19 disease may be asymptomatic. As recommended by the CDC medical personnel should be equipped with full personal protective equipment (PPE) for AGP in contact with suspected/confirmed COVID-19 patient. Therefore, it is reasonable to search for the most effective methods of intravascular access in those conditions.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest (OHCA)
* Adult ≥ 18 years old
* Non-traumatic cause of cardiac arrest

Exclusion Criteria:

* Existing do-not-attempt-resuscitation order
* OHCA patients with contraindications to IO access or IV access
* Patients with signs of obvious death, e.g. rigor mortis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Success rate of first intravascular access attempt | 1 day
  successful placement of intravascular device

SECONDARY OUTCOMES:
time to successful access | 1 day
  time to successful access
number of attempts to successful access | 1 day
  number of attempts to successful access
time to infusion | 1 day
  time to therapy including but not limited to time to fluids, antibiotics, and antiarrythmics
complication rates | 1 day
  complication rates
ROSC | 1 day
  the rate of survival to hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, PhD, Study Chair — Lazarski University
Locations (1):
- Lazarsku University, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
the investigators will decide after study finishing